CLINICAL TRIAL: NCT01973933
Title: A Open-label, Single Sequence Clinical Trial to Investigate the Pharmacokinetic/Pharmacodynamic Drug-drug Interaction of Pyrimethamine and Metformin IR After Oral Administration in Healthy Male Volunteers
Brief Title: Clinical Trial to Investigate the Pharmacokinetic/Pharmacodynamic Drug-Drug Interaction of Pyrimethamine and Metformin IR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae Yong Chung, Assistant Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPI02
Record Dates: First submitted 2013-10-27; First posted 2013-11-01 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: Metformin; Pyrimethamine; Drug interaction
MeSH Terms: interventions — Metformin; Pyrimethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin and Pyrimethamine (Experimental): Metformin 750mg(D1), Metformin 500mg(D2)/Metformin 750mg+Pyrimethamine 50mg(D7), Metformin 500mg+Pyrimethamine 50mg(D8)
  Interventions: Drug: Metformin and Pyrimethamine

INTERVENTIONS:
Drug: Metformin and Pyrimethamine
  Other Names: Diabex; Daraprim

SUMMARY:
This study aims to investigate the pharmacokinetic/pharmacodynamic drug-drug interaction of pyrimethamine and metformin IR after oral administration in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subject aged 20 to 45 at screening A body weight in the range of 50 kg (inclusive)
* 100 kg (inclusive) with ideal body weight range of +- 25% subjects who decide to participate voluntarily and write a informed consent form

Exclusion Criteria:

* subjects who have clinically significant disease of cardiovascular, respiratory, renal, endocrinological, hematological, gastrointestinal, neurological(central nervous system), psychiatric disorders or malignant tumor
* Subject judged not eligible for study participation by investigator.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
AUC(area under the plasma concentration-time curve) | Predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12h postdose
  AUC(area under the plasma concentration-time curve), Cmax(maximum plasma concentration), t1/2

SECONDARY OUTCOMES:
AUG(total area under the serum concentration-time curve for glucose) | predose and 15, 30, 45, 60, 90, 120, 150, 180min oral glucose tolerance test
  AUG (total area under the serum concentration-time curve for glucose) Gmax(maximum serum glucose concentration)

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Yong Chung, MD, PhD, Principal Investigator — Department of Clinical Pharmacology and Therapeutics, Seoul National University Bundang Hospital, Seoul, Korea
Locations (1):
- Seoul National University Bundang Hospital, Seoul, South Korea